CLINICAL TRIAL: NCT05347784
Title: Characterization of Vital Sign Circadian Fluctuations in Postsurgical Patients With or Without Complications
Brief Title: Vital Values at Circadian Markers in Postoperative Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jesper Mølgaard, MD, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: WARD-X-CIRC
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Complications; Circadian Dysrhythmia
Keywords: Postoperative physiology; Vital signs
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without postoperative complications
- Patients with postoperative complications

SUMMARY:
To describe changes in various diurnal patterns in vital values after surgery. These will be analyzed based on whether the patients have complications or no complications.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for surgery
* Expected time of surgery was more than 2 hours.
* Expected post-operative length of stay was more than 2 days.

Exclusion Criteria:

* Allergy to study materials
* Patients with a pacemaker
* Patients that were expected to be unable to cooperate with study procedures (for instance a Mini-Mental State Exam(MMSE < 25)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are drawn from two studies:
  Clinical trials registry: NCT03491137 and NCT04473001
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | From start of continuous monitoring until 12 hours after monitoring stopped.
  Any complication meeting the ICH-GCP serious adverse event(SAE) criteria:
  An SAE (...) is defined as any untoward medical occurrence that(...)
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Requires intervention to prevent permanent impairment or damage
  (May have caused a congenital anomaly/birth defect - Not relevant)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT05347784/SAP_001.pdf